CLINICAL TRIAL: NCT05333874
Title: CIPHER Study: Pilot Study to Study the Role of ctDNA in Triple Negative and HER2 Positive Early Stage Breast Cancer
Brief Title: CIPHER Study: Pilot Study to Study the Role of ctDNA in Triple Negative and HER2 Positive Early Stage
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Mridula George, MD, Assistant Professor of Medicine, Rutgers, The State University of New Jersey
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 042110; Pro2022000044 (Other: Rutgers, The State University of New Jersey)
Record Dates: First submitted 2022-04-12; First posted 2022-04-19 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Breast Cancer, Early-Onset
Keywords: Triple Negative Breast Cancer
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — Neoadjuvant Therapy; Watchful Waiting

STUDY DESIGN:
Intervention Model Description: A pilot study to evaluating the role of ctDNA in patients with Stage II-III triple negative breast cancer and HER2 positive breast cancer. Participants who have ctDNA post neoadjuvant therapy and surgery will be initiated on adjuvant systemic therapy per treating physician's choice. ctDNA will be monitored up to 24 months to study ctDNA kinetics. Signatera is intended to detect and quantify how much cancer is left in the body, to improve prognosis and help optimize treatment decisions, based on the tissue-informed testing of mutations.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Neoadjuvant chemotherapy (Active Comparator): If Circulating tumor DNA (ctDNA) blood test is positive, change in treatment can be made. Participants will be monitored with ctDNA at 60days, 3 months, 6 months, 9 months, 12 months, 18months and 24months from surgery.
  The participant's core biopsy specimens will be sent to NateraTM to sequence the primary tumor. The baseline blood work for ctDNA will be collected prior to the initiation of systemic therapy. Subsequently, ctDNA will be collected prior to each cycle of neoadjuvant chemotherapy. Participants will undergo surgery and ctDNA needs to be collected fourteen days post-surgery The treating oncologist will complete a questionnaire to determine how ctDNA impacts treatment decisions in the adjuvant setting once the results from the fourteen day ctDNA is available and at the time of ctDNA re-emergence. Participants will complete participant questionnaire at 3 months, 6months, 12months and 24 months post-operatively.
  Interventions: Drug: Neoadjuvant chemotherapy administered before surgical extraction of a tumor
- Observational (Other): Observation for triple negative breast cancer (TNBC): No adjuvant chemotherapy. Patients may complete checkpoint inhibitor from neoadjuvant setting. human epidermal growth factor receptor 2 (HER2) positive breast cancer: complete twelve months of anti-HER2 therapy, which was initiated in neoadjuvant setting), participants in the observation arm, will be monitored for Circulating tumor DNA (ct-DNA) re-emergence and systemic therapy can be added at the time of ctDNA re-emergence.
  Interventions: Other: Observational

INTERVENTIONS:
Drug: Neoadjuvant chemotherapy administered before surgical extraction of a tumor — SignateraTM is a custom-built circulating tumor DNA (ctDNA) test for treatment monitoring and molecular residual disease (MRD) assessment in patients previously diagnosed with cancer. The Signatera methodology is personalized and tumor-informed, providing each individual with a customized blood test tailored to fit the unique signature of clonal mutations found in that individual's tumor tissue. This maximizes accuracy for detecting the presence or absence of disease in a blood sample, even at levels down to a single tumor molecule in a tube of blood. Signatera is intended to detect and quantify how much cancer is left in the body, to improve prognosis and help optimize treatment decisions, based on the tissue-informed testing of mutations.
  Other Names: Neoadjuvant chemotherapy
  Arms: Neoadjuvant chemotherapy
Other: Observational — In participants, undetectable ctDNA at fourteen days will be in the observation arm (observation defined as TNBC: No adjuvant chemotherapy. Participants may complete checkpoint inhibitor from neoadjuvant setting; HER2 positive BC: Completed one year of anti-HER2 therapy from the neoadjuvant setting). No investigational drugs will be used. Samples of ctDNA will be collected at time points described in the study arm.
  Other Names: No adjuvant chemotherapy
  Arms: Observational

SUMMARY:
Primary Objective:

1) To examine the impact of Circulating tumor DNA (ctDNA) (expressed as mean tumor molecules per ml) on treatment decision making in patients with early stage breast cancer after neoadjuvant therapy and surgery

Secondary Objectives:

1. Understand ctNDA kinetics in the neoadjuvant and adjuvant setting
2. To identify any associations between clinical staging and measurable ctDNA

DETAILED DESCRIPTION:
To determine whether early detection of Circulating tumor DNA (ctDNA) after neoadjuvant systemic therapy help tailor adjuvant therapy and reduce risk of relapse in patients who are at increased risk of recurrence. Studies have shown the presence of ctDNA is associated with increased risk of relapse, it is unclear how adjuvant therapy and its effect of ctDNA impacts the risk of relapse. There is very limited data on the role of ctDNA monitoring and response to neoadjuvant/adjuvant systemic therapy in patients with human epidermal growth factor receptor 2 (HER2 ) positive breast cancer.

Natera, Inc. (NASDAQ: NTRA) has developed a minimal residual disease (MRD) assay that sequences tumor tissue to identify a unique signature of tumor mutations, then customizes a personalized PCR assay for each participant, targeting the top 16 clonal mutations found in the tumor (Signatera™). Signatera is intended to detect and quantify how much cancer is left in the body, to improve prognosis and help optimize treatment decisions, based on the tissue-informed testing of mutations.

If the ctDNA blood test is positive, change in treatment can be made after discussion with the participant and treating provider. If the decision is for observation (Observation defined for TNBC: No adjuvant chemotherapy. Participants may complete checkpoint inhibitor from neoadjuvant setting. HER2 positive breast cancer: complete 12 months of anti-HER2 therapy, which was initiated in neoadjuvant setting), participants in the observation arm, will be monitored for ct-DNA re-emergence and systemic therapy can be added at the time of ctDNA re-emergence. If the decision is made to institute systemic therapy based on the ctDNA detection, participants will be monitored with ctDNA at 60days, 3 months, 6 months, 9 months, 12 months, 18months and 24months from surgery. If ctDNA is negative, there will be no change in therapy and participants can continue on observation arm (Observation defined for TNBC: No adjuvant chemotherapy. Participants may complete checkpoint inhibitor from neoadjuvant setting. HER2 positive breast cancer: complete 12 months of anti-HER2 therapy, which was initiated in neoadjuvant setting). Participants in the observation arm will be monitored for ct-DNA re-emergence and systemic therapy can be added at the time of ctDNA re-emergence.

The treating oncologist will complete a questionnaire to determine how ctDNA impacts treatment decisions in the adjuvant setting once the results from the fourteen day ctDNA is available and at the time of ctDNA re-emergence. Participants will complete participant questionnaire at 3 months, 6months,12months and 24 months post-operatively. Participants will be followed up for five years.

ELIGIBILITY:
Inclusion Criteria:

* Participants with a diagnosis of clinical Stage II-III triple negative and/or HER2 positive breast cancer
* Age ≥ 18 years
* Estimated life expectancy of at least twelve months
* Participant must be eligible for neoadjuvant systemic therapy per treating physician
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
* Able to provide signed and dated informed consent form
* Must have ctDNA at the time of screening to be eligible for the study
* Participants enrolled on other systemic therapy trials may be eligible to participate in the study after discussion with principal investigator
* Be willing to present for medical exams and blood draws as scheduled per protocol

Exclusion Criteria:

* Evidence of metastatic breast cancer
* Any other concurrent malignancy
* Prior malignancies (except non-melanoma skin cancers, and the following in situ cancers: bladder, gastric, colon, endometrial, cervical/dysplasia, melanoma, or breast) unless a complete remission was achieved at least one year prior to study entry
* Participant is pregnant
* Serious concomitant systemic disorder that would compromise the safety of the participant or compromise the participant's ability to complete the study, at the discretion of the investigator
* Bone marrow transplant or other organ transplant recipient
* History of psychiatric illness or social situations that would limit compliance with study requirements
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2022-04-06 (Actual); Primary Completion 2027-11-28 (Estimated); Study Completion 2027-11-28 (Estimated)

PRIMARY OUTCOMES:
Detectable Circulating tumor DNA ctDNA | Five Years
  Participants with detectable ctDNA fourteen days post-operatively will have the option to change adjuvant therapy after discussion with primary provider. SignateraTM is intended to detect and quantify how much cancer is left in the body, to improve prognosis and help optimize treatment decisions, based on the tissue-informed testing of mutations.

SECONDARY OUTCOMES:
Levels of Detectable Circulating tumor DNA ctDNA | Five Years
  Participants on observation or change in adjuvant therapy will continue to be monitored with ctDNA at 60 days, 3 months, 6 months, 9 months, 12 months, 18months and 24months from surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Mridula George, MD, Principal Investigator — Rutgers Cancer Institute of New Jersey
Locations (12):
- United States (12):
  - Trinitas Hospital and Comprehensive Cancer Center, Elizabeth, New Jersey
  - RWJBarnabas Health - Robert Wood Johnson University Hospital, Hamilton, New Jersey
  - Jersey City Medical Center, Jersey City, New Jersey
  - Monmouth Medical Center - Southern Campus, Lakewood, New Jersey
  - Cooperman Barnabas Medical Center, Livingston, New Jersey
  - Monmouth Medical Center, Long Branch, New Jersey
  - Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Robert Wood Johnson Barnabas Hospital -Somerset, Somerville, New Jersey
  - Steeplechase Cancer Center, Somerville, New Jersey
  - Monmouth Medical Center Vantage Point Infusion Cente, West Long Branch, New Jersey

IPD SHARING:
Plan to Share IPD: No
The plan to share IPD will be determined by the PI and updated accordingly.

DOCUMENTS (1):
  • Informed Consent Form (2022-11-03): https://cdn.clinicaltrials.gov/large-docs/74/NCT05333874/ICF_000.pdf